CLINICAL TRIAL: NCT02280356
Title: Ultra-hypofractionated, Image-guided, Intensity-modulated Radiation Therapy in Combination With Brachytherapy for Clinically Localized, Intermediate Risk Prostate Cancer
Brief Title: Radiation Therapy in Combination With Brachytherapy for Clinically Localized, Intermediate Risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-193
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
Keywords: Radiation Therapy; Brachytherapy; 14-163
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Surveys and Questionnaires

ARMS (1):
- radiation therapy in combination with brachytherapy (Experimental): Patients will undergo low dose rate (LDR) prostate brachytherapy using Pd-103 followed approximately 4 weeks later with hypofractionated image-guided external beam radiation therapy (25Gy in 5 fractions; 5Gy x 5 fractions every other day) to the prostate & seminal vesicles. Both brachytherapy as well as external beam will be performed according to our current standards of practice using the same equipment, techniques, & treatment planning procedures. Pts will be followed post-treatment at 1, 3, 6 (+/- 4 weeks) & every 6 months (+/- 4 weeks) thereafter until 36 months. During the post-treatment followup, pts will be evaluated for urinary, bowel/rectal & sexual toxicity. Baseline measures of these domains will be obtained prior to treatment at the time of enrollment. Serum PSA levels will be drawn on the same schedule as clinical followup. Post-treatment prostate biopsies will be obtained once between 24-36 months post-treatment to evaluate pathologic response to therapy
  Interventions: Radiation: external beam radiation therapy; Radiation: brachytherapy; Behavioral: questionnaires

INTERVENTIONS:
Radiation: external beam radiation therapy
Radiation: brachytherapy
Behavioral: questionnaires
  Other Names: International Prostate Symptom Score; International Index of Erectile Function-6; EPIC urinary, bowel and sexual domain

SUMMARY:
The purpose of this study is to test the safety and side effects "of "ultra-hypofractionated" radiation therapy when used after brachytherapy (radiation implants). This treatment delivers a higher radiation dose with each treatment over a shorter period of time.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate risk prostate cancer patients will be eligible for this study. Intermediate risk grouping will be assessed per NCCN guidelines as:
* Pathologically-proven diagnosis of prostate adenocarcinoma
* PSA 10-20ng/mL or
* Gleason =7 or
* Clinical stage T2b/c
* Clinical stage T2b/c Additionally, patients will be required to meet the following criteria
* Age ≥18
* KPS≥70
* Prostate volume ≤ 60cc (cytoreductive androgen deprivation therapy prior to brachytherapy of ≤ 6 months duration will be allowed to achieve this goal). For patients with a prostate volume between 50-60ccs, hormone therapy will be at the discretion of the physician.
* International Prostate Symptom Score ≤15

Exclusion Criteria:

* Prior prostate surgery (including TURP)
* Prior history of chronic prostatitis or urethral stricture
* Inflammatory bowel disease
* Prior history of pelvic radiotherapy
* Unable to give informed consent
* Metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Kollmeier, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau (Follow Up Only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy in Combination With Brachytherapy: Patients will undergo low dose rate (LDR) prostate brachytherapy using Pd-103 followed approximately 4 weeks later with hypofractionated image-guided external beam radiation therapy to the prostate & seminal vesicles.
Period: Overall Study
Arm/Group | Radiation Therapy in Combination With Brachytherapy
Started | 45
Completed | 40
Not Completed | 5
Not completed — Not Treated | 2
Not completed — Withdrawal by Subject | 1
Not completed — Not evaluable | 2

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy in Combination With Brachytherapy
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 66 [54 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 31
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Urinary Toxicity Assessed by CTCAE v4.0
Description: Participants with Urinary Toxicity Assessed by CTCAE v4.0 at approximately 12 months of hypofractionated radiation therapy in combination with brachytherapy for the treatment of intermediate risk prostate cancer.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy in Combination With Brachytherapy
Number analyzed (Participants) | 45
Participants | 33

2. Secondary Outcome: Mean Change in International Prostate Symptom Score (IPSS) to Assess Urinary Functioning From Baseline at 12 Months
Description: The International Prostate Symptom Score/IPSS index is a seven item questionnaire that assesses urinary functioning, including urinary frequency, nocturia, weak urinary stream, hesitancy, intermittence, incomplete emptying, and urgency. Questions are rated on a six point Likert scale. Higher scores indicate more difficulty in urinary functioning. A score of 7 or less is mildly symptomatic, 8 to 19 is moderately symptomatic, and 20 to 35 is severely symptomatic. Scale range is 0-35. Total score is reported.
Time Frame: 12 months
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Radiation Therapy in Combination With Brachytherapy
Number analyzed (Participants) | 45
scores on a scale | 5 [0 to 18]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Radiation Therapy in Combination With Brachytherapy
All-Cause Mortality (participants affected / at risk) | 4/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 33/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy in Combination With Brachytherapy (N=45)
Urinary frequency (Renal and urinary disorders) | 33
Urinary urgency (Renal and urinary disorders) | 31
Erectile dysfunction (Respiratory, thoracic and mediastinal disorders) | 26
Fatigue (General disorders) | 8
Urinary incontinence (Renal and urinary disorders) | 7
Urinary tract obstruction (Renal and urinary disorders) | 6
Urinary tract pain (Renal and urinary disorders) | 6
Rectal hemorrhage (Gastrointestinal disorders) | 5
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 5
Diarrhea (Gastrointestinal disorders) | 4
Proctitis (Gastrointestinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT02280356/Prot_SAP_000.pdf